CLINICAL TRIAL: NCT06588335
Title: A Single-Center, Exploratory Study of BTLA Inhibitor (JS004) Combined with Toripalimab and Chemotherapy in the Perioperative Treatment of Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: BTLA Inhibitor (JS004) Combined with Toripalimab and Chemotherapy in the Perioperative Treatment of Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanPPH-WEILI
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab; TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- S004+ Toripalimb+Chemotherapy (paclitaxel + cisplatin) (Experimental): Neoadjuvant therapy stage: JS004+ triplizumab + chemotherapy (paclitaxel + cisplatin), 2 cycles; Operation stage: Surgery 3-8 weeks after the last neoadjuvant; Postoperative maintenance treatment stage: Maintenance therapy was started at 4 weeks ±7 days after surgery. Postoperative maintenance therapy should be initiated no later than 10 weeks after surgery.
  Interventions: Drug: BTLA inhibitor (JS004); Drug: Toripalimab; Drug: Paclitaxel, Cisplatin

INTERVENTIONS:
Drug: BTLA inhibitor (JS004) — BTLA inhibitor (JS004):200mg, intravenous infusion , d1, Q3W;
Drug: Toripalimab — Toripalimab:240mg,intravenous infusion, d1, Q3W;
Drug: Paclitaxel, Cisplatin — Paclitaxel, 175mg/m2, intravenous infusion, d1, Q3W; Cisplatin, 75mg/m2, intravenous infusion, d1, Q3W;

SUMMARY:
This is a single-center, single-arm, phase II study, aiming to preliminarily explore the efficacy and safety of JS004 combined with toripalimab and chemotherapy for perioperative treatment of locally advanced thoracic esophageal squamous cell carcinoma that is resectable. The plan is to enroll 20 patients with locally advanced resectable thoracic esophageal cancer. In the neoadjuvant treatment phase, patients will receive JS004 + toripalimab + chemotherapy (paclitaxel + cisplatin) for 2 cycles. This will be followed by the surgical phase: surgery will be performed 3-8 weeks after the last dose of neoadjuvant treatment. In the postoperative maintenance treatment phase, maintenance treatment will start 4 weeks ± 7 days after surgery, but no later than 10 weeks after surgery. For patients with R0 resection confirmed by postoperative pathology, they will receive maintenance treatment with JS004 + toripalimab for up to 15 cycles. For patients with non-R0 resection, they will receive maintenance treatment with JS004 + toripalimab combined with standard radiation or chemotherapy (selected by the investigator based on esophageal cancer guidelines). During the study, the maximum number of cycles of JS004 combined with toripalimab is 17 cycles (approximately 1 year).

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participates in this study, signs the informed consent form, has good compliance, and cooperates with the follow-up;
2. Age 18-75 years old, including 18 and 75 years old, both male and female;
3. Histologically or cytologically confirmed clinical stage of locally advanced (T1N1-3M0 or T2-3N0-3M0) thoracic esophageal squamous cell carcinoma (8th UICC-TNM staging);
4. Enhanced CT of the neck shows no suspicious metastatic lymph nodes (excluding lymph nodes in the esophageal cancer area), and imaging examination shows no distant metastasis;
5. ECOG: 0~1 score;
6. Expected to achieve R0 resection;
7. No previous anti-tumor treatment for esophageal cancer, including chemotherapy, radiotherapy (including planned radiotherapy during the study period), hormone therapy and immunotherapy;
8. Have measurable lesions or assessable non-measurable lesions (according to RECIST 1.1 criteria);
9. The function of important organs meets the following requirements (no use of any blood components and cell growth factors is allowed within 2 weeks before the screening examination): a. Absolute neutrophil count (ANC) ≥1.5×10^9/L; b. Platelets ≥100×10^9/L; c. Hemoglobin ≥90g/dL; d. Serum albumin ≥2.8g/dL; e. Total bilirubin ≤1.5×ULN, ALT, AST and/or AKP ≤2.5×ULN; f. Serum creatinine ≤1.5×ULN or creatinine clearance ≥60mL/min (calculated by Cockcroft-Gault formula); g. International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN (for those using a stable dose of anticoagulant therapy such as low molecular weight heparin or warfarin, and the INR is within the expected therapeutic range of the anticoagulant, they can be screened);
10. For female subjects of childbearing potential, a urine or serum pregnancy test must be performed within 72 hours prior to receiving the first study drug, and the result must be negative, and they are willing to use effective contraception during the study period and for 6 months after the last dose.

Exclusion Criteria:

1. Patients at high risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation.
2. Patients with uncontrolled, recurrent pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
3. Patients with severe dysfunction of the heart, lung, liver, kidney, hematopoietic system, endocrine system, or cachexia.
4. Patients who have received any of the following treatments: a. Major surgery (except for diagnostic tissue biopsy) or serious trauma within 4 weeks prior to first study drug administration. b. Anti-cancer therapy (including chemotherapy, radiotherapy, immunotherapy, targeted therapy, biotherapy, or tumor embolization) within 4 weeks prior to first study drug administration. c. Any investigational drug within 4 weeks prior to first study drug administration. d. Anti-cancer vaccine or live vaccine within 4 weeks prior to first study drug administration. e. Systemic corticosteroid therapy (>10 mg prednisone equivalent per day) or other immunosuppressants within 2 weeks prior to first study drug administration, except for local inflammation of the esophagus and prevention of allergy and nausea/vomiting.
5. Patients whose previous anti-cancer therapy toxicity has not recovered to ≤CTCAE Grade 1 (except for alopecia).
6. Patients with sodium, potassium, or calcium laboratory abnormalities >Grade 1 that cannot be corrected within 2 weeks prior to first study drug administration.
7. Patients with any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonitis, uveitis, colitis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism), except for vitiligo or childhood asthma/allergy that has resolved without the need for intervention in adulthood.
8. Patients with a history of immunodeficiency, including HIV-positive, other acquired or congenital immunodeficiency disorders, organ transplant, or allogeneic bone marrow transplant.
9. Patients with uncontrolled cardiac conditions, such as (1) NYHA Class II or higher heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, or (4) clinically significant arrhythmias requiring intervention.
10. Patients with a serious infection (CTCAE >Grade 2) within 4 weeks prior to first study drug administration, active lung inflammation on baseline imaging, or symptoms/signs of infection within 2 weeks prior to first study drug administration requiring oral or IV antibiotics (except for prophylactic use).
11. Patients with active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL) or active hepatitis C (positive HCV antibody and detectable HCV-RNA).
12. Patients with known hypersensitivity, allergy, or contraindication to JS004, toripalimab, or any of their formulation components.
13. Patients with any other malignancy, except for low-risk malignancies (5-year survival rate >90%) such as fully treated basal cell or squamous cell skin cancer or cervical carcinoma in situ.
14. Pregnant or breastfeeding women, or patients of reproductive potential unwilling or unable to use effective contraception.

The investigator may also exclude patients if there are other factors that may lead to premature discontinuation from the study, such as other serious concurrent illnesses (including psychiatric disorders) requiring concomitant treatment, high risk of recurrence of recent serious illness (e.g., myocardial infarction, stroke), severe laboratory abnormalities, or family/social factors that may affect patient safety or data collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | up to 3 weeks after neoadjuvant
  pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.assessment criteria after neoadjuvant therapy, as defined by the CAP (College of American Pathologists) and NCCN (National Comprehensive Cancer Network) guidelines.

SECONDARY OUTCOMES:
Major pathological response rate (MPR) | up to 3 weeks after neoadjuvant
  mPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes in neoadjuvant therapy
Event-free lifetime (EFS) | up to 3 years
  EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause. EFS determined either by biopsy assessed by central pathologist or by imaging using RECIST 1.1 assessed by investigator
Overall survival (OS) | up to 3 years
  OS is defined as the time from randomization until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: LI WEI, Principal Investigator — Henan Provincial People&#39;s Hospital

IPD SHARING:
Plan to Share IPD: No